CLINICAL TRIAL: NCT05986461
Title: Spatially Resolved Transcriptomics Reveals Phenotype-specific Molecular Signatures in Complex Regional Pain Syndrome
Brief Title: Spatially Transcriptomics Reveals Molecular Signatures in CRPS
Status: Recruiting | Type: Observational
Sponsor: Seoul National University (Other)
Collaborators: Hanyang University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Professor, Seoul National University
Other Study IDs: 2304-052-1421
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples With DNA — Punch biopsied skin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to understand phenotype-specific molecular signatures in patients with complex regional pain syndrome (CRPS).

DETAILED DESCRIPTION:
Participants who meet the diagnostic criteria for CRPS, aged 19~80 years, and agree to participate in this study will undergo a 4mm-sized skin punch biopsy in the involved limb, as well as the contralateral side (internal control).

Spatial transcriptomics will be used to identify immune cell signatures and differentially regulated genes (DEGs) in the epidermis, vasculature, sweat gland, and nerve plexus of the involved ipsilateral (vs contralateral) side of the patient's skin.

ELIGIBILITY:
Inclusion Criteria:

* Meets the Budapest diagnostic criteria
* Consents to participation in this study
* Aged between 19 and 80 years old
* Symptoms and/or signs of sensory, vasomotor, and sudomotor changes

Exclusion Criteria:

* Who do not agree to participate in this study
* Who has contraindications for skin punch biopsy (e.g. thrombocytopenia, taking anticoagulant drugs)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CRPS
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | At the time of biopsy
  Intensity of pain (now, weekly avarege, weekly maximum)
Thermography | At the time of diagnosis
  Thermography of the involved limb
Quantitative Sensory Testing (QST) | At the time of diagnosis
  Vibration Detection Threshold (VDT), Cold Detection Threshold (CDT)

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youn Moon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taylor SS, Noor N, Urits I, Paladini A, Sadhu MS, Gibb C, Carlson T, Myrcik D, Varrassi G, Viswanath O. Complex Regional Pain Syndrome: A Comprehensive Review. Pain Ther. 2021 Dec;10(2):875-892. doi: 10.1007/s40122-021-00279-4. Epub 2021 Jun 24. PMID 34165690
- [Result] Rao A, Barkley D, Franca GS, Yanai I. Exploring tissue architecture using spatial transcriptomics. Nature. 2021 Aug;596(7871):211-220. doi: 10.1038/s41586-021-03634-9. Epub 2021 Aug 11. PMID 34381231
- [Result] Birklein F, Drummond PD, Li W, Schlereth T, Albrecht N, Finch PM, Dawson LF, Clark JD, Kingery WS. Activation of cutaneous immune responses in complex regional pain syndrome. J Pain. 2014 May;15(5):485-95. doi: 10.1016/j.jpain.2014.01.490. Epub 2014 Jan 23. PMID 24462502
- [Result] Escolano-Lozano F, Gries E, Schlereth T, Dimova V, Baka P, Vlckova E, Konig S, Birklein F. Local and Systemic Expression Pattern of MMP-2 and MMP-9 in Complex Regional Pain Syndrome. J Pain. 2021 Oct;22(10):1294-1302. doi: 10.1016/j.jpain.2021.04.002. Epub 2021 Apr 20. PMID 33892152
- [Result] Stahl PL, Salmen F, Vickovic S, Lundmark A, Navarro JF, Magnusson J, Giacomello S, Asp M, Westholm JO, Huss M, Mollbrink A, Linnarsson S, Codeluppi S, Borg A, Ponten F, Costea PI, Sahlen P, Mulder J, Bergmann O, Lundeberg J, Frisen J. Visualization and analysis of gene expression in tissue sections by spatial transcriptomics. Science. 2016 Jul 1;353(6294):78-82. doi: 10.1126/science.aaf2403. PMID 27365449
- [Result] Ji AL, Rubin AJ, Thrane K, Jiang S, Reynolds DL, Meyers RM, Guo MG, George BM, Mollbrink A, Bergenstrahle J, Larsson L, Bai Y, Zhu B, Bhaduri A, Meyers JM, Rovira-Clave X, Hollmig ST, Aasi SZ, Nolan GP, Lundeberg J, Khavari PA. Multimodal Analysis of Composition and Spatial Architecture in Human Squamous Cell Carcinoma. Cell. 2020 Jul 23;182(2):497-514.e22. doi: 10.1016/j.cell.2020.05.039. Epub 2020 Jun 23. PMID 32579974
- [Result] Andronic D, Andronic O, Juengel A, Berli MC, Distler O, Brunner F. Skin biomarkers associated with complex regional pain syndrome (CRPS) Type I: a systematic review. Rheumatol Int. 2022 Jun;42(6):937-947. doi: 10.1007/s00296-021-05061-5. Epub 2022 Jan 8. PMID 34997300